CLINICAL TRIAL: NCT00677794
Title: Small Bowel Cleansing Prior to Video Capsule Endoscopy Examination: a Randomized, Blinded, Controlled Trial
Brief Title: Small Bowel Cleansing Prior to Video Capsule Endoscopy Examination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: small bowel cleansing and VCE
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Endoscopy
Keywords: Video Capsule Endoscopy; Small Bowel
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Clear fluids only after lunch.
  Interventions: Drug: Clear fluids
- 2 (Active Comparator): Two sachets of picosalax the evening prior to Video Capsule Endoscopy (VCE).
  Interventions: Drug: Picosalax
- 3 (Active Comparator): Polyethylene glycol, 2 liters the evening prior to Video Capsule Endoscopy (VCE).
  Interventions: Drug: Polyethylene glycol

INTERVENTIONS:
Drug: Clear fluids — Clear fluids only after lunch.
  Arms: 1
Drug: Picosalax — Two sachets the evening prior to Video Capsule Endoscopy (VCE).
  Arms: 2
Drug: Polyethylene glycol — Two (2) litres the evening prior to Video Capsule Endoscopy (VCE).
  Arms: 3

SUMMARY:
There remains debate regarding whether small bowel cleansing is required prior to video capsule endoscopy, and if so, which method is best. This study prospectively tests cleansing with no preparation, preparation with picosalax, and preparation with polyethylene glycol.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing VCE.

Exclusion Criteria:

* bowel obstruction or ileus;
* known stricture or fistula;
* previous small bowel surgery;
* severe gastroparesis or motility disorder
* renal impairment (serum creatinine over normal range within three months of study);
* congestive heart failure;
* cirrhosis;
* implanted cardiac pacemaker or defibrillator or other electromedical device;
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2008-03; Primary Completion 2013-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
small bowel cleansing | during exam

SECONDARY OUTCOMES:
yield of Video Capsule Endoscopy (VCE) in iron deficiency | during study
tolerance of preparation | during preparation
effect of preparation on blood chemistry | 24 hours after ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Hookey L, Louw J, Wiepjes M, Rubinger N, Van Weyenberg S, Day AG, Paterson W. Lack of benefit of active preparation compared with a clear fluid-only diet in small-bowel visualization for video capsule endoscopy: results of a randomized, blinded, controlled trial. Gastrointest Endosc. 2017 Jan;85(1):187-193. doi: 10.1016/j.gie.2016.07.028. Epub 2016 Jul 21. PMID 27451294